CLINICAL TRIAL: NCT00734747
Title: Evaluation of the Medigus SRS Endoscopic Stapling System for the Treatment of Gastro-Esophageal Reflux Disease (GERD)
Brief Title: Safety and Efficacy the Medigus SRS Endoscopic Stapling System in Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aviel Roy-Shapira, M.D. (Industry)
Responsible Party: Sponsor-Investigator, Aviel Roy-Shapira, M.D., Study director, Medigus Ltd
Organization: Medigus Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCLP09002
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; Gastroesophageal Reflux; Fundoplication; Endoluminal; Gastroesophageal Flap Valve
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medigus SRS Endoscopic Stapling System (Experimental): Endoluminal fundoplication for the treatment of GERD
  Interventions: Device: Medigus SRS endoscopic stapling system

INTERVENTIONS:
Device: Medigus SRS endoscopic stapling system — The system is designed to staple the stomach to the esophagus in 2 or 3 locations using a quintuplet of standard B shaped, 4.8 mm titanium staples in each location.
  Other Names: endoluminal treatment of GERD; Incisionless treatment of GERD

SUMMARY:
The study is designed to test the safety and efficacy of the Medigus SRS endoscopic stapling system for the treatment of GERD.

The system allows the operator to staple the stomach to the esophagus,in order to restore the gastroesophageal flap valve. The effect of the stapling is similar to a common operation for GERD (partial fundoplication) but is done through the mouth, and incision into the abdomen is not needed.

The hypothesis of the study is that the treatment will be effective in improving GERD related quality of life by 50% or more in the majority of the subjects, and that the procedure will be as safe as surgery.

ELIGIBILITY:
Inclusion Criteria:

* History of GERD related symptoms for at least 2 years.
* Recent objective evidence of GERD, demonstrated by a 24h pH acid exposure test.
* History of daily intake of proton pump inhibitors (PPIs) for at least 6 months, with significant relief of symptoms (i.e., difference in GERD Health Related Quality of Life (GERD HRQL) scores on and off PPI > =6).
* GERD-HRQL ≥20 off of PPI's

Exclusion Criteria:

* Hiatal hernia > 3 cm or a paraesophageal hernia
* Barrett's esophagus or grade IV esophagitis
* Esophageal stricture, ring or web causing symptoms of dysphagia
* Grade I Flap valve according Hill's classification
* History of co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aviel Roy-Shapira, M.D., Study Director — Medigus Ltd
Locations (6):
- United States (2):
  - UC San Diego, San Diego, California
  - Indiana University Hospital, Indianapolis, Indiana
- Akh Vienna City General Hospital, Vienna, Austria
- Med.Klinik Universitatsmedizin, Mainz, Germany
- Deenanath Mangeshkar Hospital and Medical Research Center, Pune, India
- Medical University of Milan - San Donato Hospital, Milan, Italy

REFERENCES:
- [Result] Zacherl J, Roy-Shapira A, Bonavina L, Bapaye A, Kiesslich R, Schoppmann SF, Kessler WR, Selzer DJ, Broderick RC, Lehman GA, Horgan S. Endoscopic anterior fundoplication with the Medigus Ultrasonic Surgical Endostapler (MUSE) for gastroesophageal reflux disease: 6-month results from a multi-center prospective trial. Surg Endosc. 2015 Jan;29(1):220-9. doi: 10.1007/s00464-014-3731-3. Epub 2014 Aug 19. PMID 25135443
- [Result] Kim HJ, Kwon CI, Kessler WR, Selzer DJ, McNulty G, Bapaye A, Bonavina L, Lehman GA. Long-term follow-up results of endoscopic treatment of gastroesophageal reflux disease with the MUSE endoscopic stapling device. Surg Endosc. 2016 Aug;30(8):3402-8. doi: 10.1007/s00464-015-4622-y. Epub 2015 Nov 4. PMID 26537905

RESULTS

PARTICIPANT FLOW:
Period: SRS Procedure
Arm/Group | Medigus SRS Endoscopic Stapling System
Started | 72
Completed | 69
Not Completed | 3
Not completed — No staples placed | 3
Period: 6 Month Follow-up
Arm/Group | Medigus SRS Endoscopic Stapling System
Started | 69
Completed | 66
Not Completed | 3
Not completed — Did not meet inclusion criteria | 3

BASELINE CHARACTERISTICS:
Population: All subjects consented for enrollment
Arm/Group | Medigus SRS Endoscopic Stapling System
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] | 47.5 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Region of Enrollment [Number; unit: participants]
  Austria | 9
  United States | 38
  Italy | 5
  Germany | 7
  India | 13
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 26.5 (4.3)
GERD HRQL on PPI [Median (Standard Deviation); unit: units on a scale] — Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) questionnaire, also known as Velanovich score. The questionnaire consists of 10 questions with responses of 0-5. The responses of the 10 questions are totaled (range of 0-50) where a higher total indicates more severe disease than a lower total. This questionnaire was administered while the subjects were taking proton pump inhibitor (PPI) medication.
  units on a scale | 15 (7.5)
GERD HRQL off PPI [Median (Standard Deviation); unit: units on a scale] — Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) questionnaire, also known as Velanovich score. The questionnaire consists of 10 questions with responses of 0-5. The responses of the 10 questions are totaled (range of 0-50) where a higher total indicates more severe disease than a lower total. This questionnaire was administered while the subjects were not taking proton pump inhibitor (PPI) medication (i.e. off-PPI)
  units on a scale | 29 (6.2)
% total time pH < 4 [Mean (Standard Deviation); unit: % total time] — Ambulatory, 24 hour esophageal pH measurement; Baseline value calculated for n=66 participants evaluated at 6 months.
  % total time | 10.9 (10.7)
Hill Grade [Number; unit: participants] — Hill Scores indicating the status of the patients' Gastroesophageal Flap Valve (GEFV). A satisfactory flap valve has a Hill Grade of 1 or 2.
  participants
    Hill Grade <= 2 | 22
    Hill Grade >=2 | 43
    No baseline measurement | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With >= 50% Improvement in GERD Health Related Quality of Life (GERD-HRQL - Velanovich) Score
Description: Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) questionnaire, also known as Velanovich score. The questionnaire consists of 10 questions with responses of 0-5. The responses of the 10 questions are totaled (range of 0-50) where a higher total indicates more severe disease than a lower total. This questionnaire was administered while the subjects were not taking proton pump inhibitor (PPI) medication (i.e. off-PPI). Criterion for success was an improvement >= 50% compared to baseline, at six months post procedure in at least 53% of the subjects (53% is the lower boundary of the 95% confidence interval)
Time Frame: Six months
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Arm/Group | Medigus SRS Endoscopic Stapling System
Number analyzed (Participants) | 66
percentage of total participants | 73 [60 to 83]

2. Primary Outcome: Serious Adverse Events (SAEs)
Description: The primary safety endpoint consisted of all treatment-related adverse events, during and after the SRS procedure. The primary safety endpoint consisted of all treatment-related adverse events, during and after the SRS procedure. "Treatment-related" events were conventionally defined as those which occurred in the first 30 days post-procedure. The SAEs presented here include all SAEs from the study, including one that occurred 35 days post-procedure (suicidal behavior). There was an interim review of early Serious Adverse Events (SAEs) after the first 24 patients. Protocol and device changes were then implemented, prior to the final 48 patients. Therefore, the SAEs are presented in two categories consisting of the first 24 patients and the final 48 patients.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Medigus SRS Endoscopic Stapling System
Number analyzed (Participants) | 72
participants
  Serious Adverse Event - First 24 patients | 8
  Serious Adverse Events - final 48 participants | 2

3. Secondary Outcome: Reduction of Acid Exposure (%Time pH<4) on Off PPI Ambulatory 24h Acid Exposure Test
Description: Esophageal pH (off PPI therapy) was measured in 66 patients pre-procedure and 64 patients at 6 months post-procedure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of time pH <4.0
Arm/Group | Medigus SRS Endoscopic Stapling System
Number analyzed (Participants) | 64
percentage of time pH <4.0 | 7.3 (5.1)
Statistical Analysis 1: Comparison: Medigus SRS Endoscopic Stapling System; Test type: Superiority or Other; p < .001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Reduction of Proton Pump Inhibitor (PPI) Use, as Reported by Subject
Time Frame: 6 months
Population: Note: 1 of the 66 participants was not taking proton pump inhibitors (PPIs) at baseline, therefore they were excluded from the analysis of PPI use reduction.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Medigus SRS Endoscopic Stapling System
Number analyzed (Participants) | 65
percentage of subjects
  % patients who eliminated PPI use | 65 [52 to 76]
  % patients who reduced PPI use by >50% | 85 [72 to 92]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Medigus SRS Endoscopic Stapling System
Serious Adverse Events (participants affected / at risk) | 10/72
Other Adverse Events (participants affected / at risk) | 43/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medigus SRS Endoscopic Stapling System (N=72)
Upper GI bleed (Gastrointestinal disorders) | 1 (1)
Pain and fever (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 1 (1)
Suicidal behavior (Psychiatric disorders) | 1 (1)
Pleural effusion, esophageal leak (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax/pneumoperitoneum (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medigus SRS Endoscopic Stapling System (N=72)
Increase belching (Gastrointestinal disorders) | 4 (4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less